CLINICAL TRIAL: NCT02358304
Title: Treatment of Aggressive Central Giant Cell Granuloma
Brief Title: Efficacy of Nasal Spray Calcitonin on Recurrence of Aggressive Central Giant Cell Granuloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Tabrizi, Assistant professor of Shiraz University of Medical Sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1234567
Record Dates: First submitted 2015-01-16; First posted 2015-02-06 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Central Giant Cell Granuloma
MeSH Terms: conditions — Granuloma, Giant Cell

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a:Patients with aggressive CGCG (Active Comparator): Patients had been clinically with CGCG and confirmed by histopathological findings were selected for the study. Gender, age, medical history, symptoms, size, and site of the lesions , duration of disease were recorded. Local ethical committee approval was obtained before the trial started and all patients gave written informed consent. Patients were randomly divided into two groups .First group received nasal spray calcitonin 200 IU/ day for 3 months after surgical curettage was done.
  Interventions: Drug: nasal spray calcitonin
- b; Patients with aggressive CGCG (Placebo Comparator): Patients had been clinically with CGCG and confirmed by histopathological findings were selected for the study. Gender, age, medical history, symptoms, size, and site of the lesions , duration of disease were recorded. Local ethical committee approval was obtained before the trial started and all patients gave written informed consent. Patients were randomly divided into two groups . second group received placebo after surgical curettage for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: nasal spray calcitonin — recurrence rate of aggressive CGCG will be recorded after the use of nasal spray calcitonin
  Arms: a:Patients with aggressive CGCG
Drug: Placebo
  Arms: b; Patients with aggressive CGCG

SUMMARY:
The main objective of this randomised clinical trial is to is to compare the frequency of recurrence between patients who received nasal spray calcitonin after curettage of Central Giant Cell Granuloma and without it.

DETAILED DESCRIPTION:
A total of 24 patients with aggressive Central Giant Cell Granuloma (CGCG )will be selected . All examinations were performed by calibrated clinicians and gender, age, medical history, symptoms, lesion size and site, disease duration and form of treatment were recorded for all participant. Radiographic examination with cone beam computed tomography (CBCT) and panoramic radiograph was done for all patients. All patients were randomly assigned to one of two treatment groups; 2 weeks after the biopsies were taken.

The case group (n =12 with) underwent 200 IU/day ones a day for 3 months after the surgeries. conservative curettage surgical procedure was done for them. while placebo was treated by curettage of CGCGs and received a placebo ones a day for 3 months after surgeries.. Patients were followed up by a maxillofacial surgeon who did not participated in surgeries.None of surgeons did not aware about the research before and during the operations.Patients were blinded from the drugs which they received after surgeries.

All patients were follow up for 5 years after operations. Recurrence lesions were documented by clinical and radiographical examinations and proved by histopathological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* clinical and histopathological diagnosis of aggressive CGCG based on accepted criteria established by chuong etal normal level of calcitonin and serum Parathyroid hormone(PTH) Patients of both sexes between 13 to 30 year's old Patients who gave written informed consent Patients who were willing for evaluation in the fallow up session Primary size of the lesion should be more than 5 cm in CBCT

Exclusion Criteria:

* Participants demonstrating a systemic disease which affects bone healing,brown tumor ,pregnancy , recently corticosteroid therapy , previous surgical intervention for CGCG or refused study enrollment and whom they could not continue the study for private or social reasons were excluded from the study sample.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Relief sign &symptom and clinical features | 5 years

SECONDARY OUTCOMES:
recurrence rate of CGCG | 5 years
  Recurrence lesions were documented by clinical and radiographical examinations and proved by histopathological evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: touba karagah, DMD, Principal Investigator — Shiraz University of Medical Sciences; Sorena Fardisi, DMD, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz university of medical sciences, Shiraz, Fars, Iran